CLINICAL TRIAL: NCT00180934
Title: Interest of a Reirradiation With Concomitant Chemotherapy After Salvage Surgery for Recurrence of Head and Neck Cancer in Irradiated Area: a Multicentric Phase III Randomized Trial
Brief Title: Reirradiation With Concomitant Chemotherapy After Salvage Surgery for Recurrence of Head and Neck Cancer in Irradiated Area
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: JANORL; CSET 98/656
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2005-12-23 (Estimated); Status verified 2005-09

CONDITIONS: Recurrence of Head and Cancer in Irraiated Area
MeSH Terms: interventions — Re-Irradiation

INTERVENTIONS:
Procedure: Reirradiation with concomitant chemotherapy

SUMMARY:
Interest of a reirradiation with concomitant chemotherapy after salvage surgery for recurrence of head and cancer in irradiated area : a multicentric Phase III randomized trial

ELIGIBILITY:
Inclusion Criteria:

* head and neck squamous cancer
* both sexes
* >=18 years
* recurrence treated by surgery and initially treated by radiotherapy
* with written informed consent at entry time

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280
Dates: Start 1999-07

PRIMARY OUTCOMES:
Overall survival at 3 years

SECONDARY OUTCOMES:
Local event-free survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: François JANOT, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France